CLINICAL TRIAL: NCT00022178
Title: An Open Label Prospective Randomised Study Comparing The Use Of Vincristine, Adriamycin And Cyclophosphamide (VAC) Versus Epirubicin, Cisplatin And Continuous 5-Flourouracil (ECF) In Patients With Unknown Primary Carcinoma (UPC)
Brief Title: Combination Chemotherapy in Treating Patients With Metastatic Cancer of an Unknown Site of Origin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068792; CHNT-VAC-VS-ECF; EU-20041
Record Dates: First submitted 2001-08-10; First posted 2004-02-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2002-02

CONDITIONS: Carcinoma of Unknown Primary
Keywords: adenocarcinoma of unknown primary; squamous cell carcinoma of unknown primary; undifferentiated carcinoma of unknown primary; newly diagnosed carcinoma of unknown primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — Cisplatin; Cyclophosphamide; Doxorubicin; Epirubicin; Fluorouracil; Vincristine

INTERVENTIONS:
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: epirubicin hydrochloride
Drug: fluorouracil
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective for metastatic cancer of an unknown site of origin.

PURPOSE: Randomized phase III trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have metastatic cancer of an unknown site of origin.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of the regimens, in terms of tumor response, progression-free survival, and overall survival of vincristine, doxorubicin, and cyclophosphamide vs epirubicin, cisplatin, and fluorouracil in patients with metastatic carcinoma of unknown primary. II. Compare the toxicity of these regimens in these patients. III. Compare quality of life and symptom control in patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to presence of liver metastases (yes vs no) and type of tumor (adenocarcinoma vs non-adenocarcinoma). Patients are randomized to one of two treatment arms. Arm I: Patients receive vincristine IV, doxorubicin IV, and cyclophosphamide IV on day 1. Arm II: Patients receive epirubicin IV and cisplatin IV over 4 hours on day 1 and fluorouracil IV continuously on days 1-21. Treatment in both arms repeats every 3 weeks for 3-6 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, at the end of courses 2, 4, and 6, and 1 month after completion of therapy. Patients are followed at 1 month and then until death.

PROJECTED ACCRUAL: A total of 398 patients (199 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic carcinoma of unknown primary Adenocarcinoma or non-adenocarcinoma No axillary lymph node metastases as sole site of disease in female patients No peritoneal carcinomatosis as sole site of disease in female patients No squamous cell carcinoma in cervical lymph nodes as sole site of disease in male or female patients No neuroendocrine tumors No elevated alpha-fetoprotein, beta-HCG, or PSA

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin less than 1.8 mg/dL Renal: Creatinine less than 1.5 times upper limit of normal (ULN) Urea less than 1.5 times ULN Glomerular filtration rate at least 60 mL/min Cardiovascular: LVEF at least 50% by echocardiogram or MUGA scan No uncontrolled angina pectoris No heart failure No clinically significant uncontrolled cardiac arrhythmias No abnormal EKG Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 1 year after study No other prior malignancy except adequately treated non-melanoma skin cancer or carcinoma in situ of the cervix No medical or psychiatric condition that would preclude study No other serious uncontrolled medical condition

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for carcinoma of unknown primary Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed except to sole site of measurable or evaluable disease Concurrent palliative radiotherapy allowed except to sole site of measurable or evaluable disease Surgery: Not specified Other: No other concurrent experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Juan W. Valle, MD, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom